CLINICAL TRIAL: NCT00879749
Title: A Phase I Study to Determine Safety, Tolerability and Bioactivity of Nexvax2 in HLA DQ2+ Volunteers With Coeliac Disease Following a Long-term, Strict Gluten-free Diet
Brief Title: Safety Study of Nexvax2 in Subjects With Coeliac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nexpep Pty Ltd (Industry)
Responsible Party: Robert Anderson/Chief Executive Officer, Nexpep Pty Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nexvax2-001
Record Dates: First submitted 2009-04-08; First posted 2009-04-10 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Coeliac Disease; Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Other: Placebo
- Nexvax2 (Experimental)
  Interventions: Biological: 9 micrograms Nexvax2; Biological: 30 micrograms Nexvax2; Biological: 90 micrograms Nexvax2; Biological: 60 micrograms Nexvax2; Biological: Up to 900 micrograms Nexvax2

INTERVENTIONS:
Biological: 9 micrograms Nexvax2 — 9 micrograms, weekly intra-dermal injection, 3 week duration
  Arms: Nexvax2
Biological: 30 micrograms Nexvax2 — 30 micrograms, weekly intra-dermal injection, 3 week duration
  Arms: Nexvax2
Biological: 90 micrograms Nexvax2 — 90 micrograms, weekly intra-dermal injection, 3 week duration
  Arms: Nexvax2
Biological: 60 micrograms Nexvax2 — 60 micrograms, weekly intra-dermal injection, 3 week duration
  Arms: Nexvax2
Biological: Up to 900 micrograms Nexvax2 — Up to 900 micrograms, weekly intra-dermal injection, 3 week duration
  Arms: Nexvax2
Other: Placebo — 100 microlitres 0.9% sterile sodium chloride for injection
  Arms: Saline

SUMMARY:
The main purpose of this study is to determine the safety of weekly injections of Nexvax2 given for three weeks to patients with coeliac disease who have been on a gluten-free diet.

The second purpose of this study is to compare the immune response over the three week study period in coeliac disease patients given Nexvax2 compared to those given saline.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18 to 60 years (inclusive)
2. Have coeliac disease meeting the following criteria:

   * the Principal Investigator is satisfied coeliac disease has been correctly diagnosed,
   * HLA DQ2 genotype (both HLA DQA1*05 and DQB1*02, homo- or hetero-zygous),
   * no known or suspected gluten exposure for 2 months prior to enrolment
   * were prescribed and have intended to follow a gluten-free diet for at least one year
   * antibodies to tissue transglutaminase (tTG) IgA and/or deamidated gliadin peptide (DGP) IgA and IgG within normal reference range at time of screening.
3. Either male or non-lactating, non-pregnant females who are postmenopausal, sterile or using at least two acceptable and highly effective birth control methods.

Key Exclusion Criteria:

1. Subjects possess the genes encoding HLA DQ8 (either DQA1*03 or DQB1*0302).
2. Uncontrolled complications of coeliac disease which, in the opinion of the Investigator, would impact immune response or pose an increased risk to the subject.
3. Systemic biological agents less than 6 months prior to Day 1.
4. Receipt of systemic immunomodulatory agents or experimental drugs less than 30 days prior to Day 1.
5. Any of the following laboratory abnormalities at Screening:

   * ALT, AST or alkaline phosphatase (ALP) > 1.5 times the upper limit of normal (ULN)
   * Calculated creatinine clearance < 80 mL/min
   * Haemoglobin (Hb) outside of the normal range
   * Platelet count <125 x 109/L
   * Serum potassium outside of the normal range
   * White blood cell (WBC) count outside of the normal range
   * Thyroid stimulating hormone (TSH) outside of the normal range
   * Any other clinically significant abnormal lab values, as determined by the Clinical Investigator.
6. Subjects who smoke or who have smoked at all in the past 3 months.
7. Positive pregnancy test at Screening or Baseline.
8. History of any medically significant condition considered by the Investigator to adversely affect participation in the trial.
9. Non-compliance with a gluten free diet or flare in coeliac disease symptoms from Screening to Baseline.
10. Clinically relevant abnormality on ECGs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Brown, MBBS PhD FRACP, Principal Investigator — The Alfred Hospital, Victoria; James Daveson, MBBS FRACP, Principal Investigator — Princess Alexandra Hospital, Queensland
Locations (2):
- Australia (2):
  - Q-Pharm Pty Ltd, Herston, Queensland
  - Nucleus Network - Centre for Clinical Studies, Melbourne, Victoria

REFERENCES:
- [Derived] Tye-Din JA, Stewart JA, Dromey JA, Beissbarth T, van Heel DA, Tatham A, Henderson K, Mannering SI, Gianfrani C, Jewell DP, Hill AV, McCluskey J, Rossjohn J, Anderson RP. Comprehensive, quantitative mapping of T cell epitopes in gluten in celiac disease. Sci Transl Med. 2010 Jul 21;2(41):41ra51. doi: 10.1126/scitranslmed.3001012. PMID 20650871